CLINICAL TRIAL: NCT02766166
Title: Critical Health Assessment and Outcomes Score/Study
Acronym: CHAOS
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Cincinnati (Other); Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: CR02_2017-5045 (central IRB)
Record Dates: First submitted 2016-05-02; First posted 2016-05-09 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Critical Illness; Death, Sudden
MeSH Terms: conditions — Critical Illness; Death, Sudden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Predictive Monitoring
- No Predictive Monitoring

SUMMARY:
CHAOS is based on the investigator's new and exciting results from pre-clinical and large longitudinal multi-center observational clinical studies of critically ill patients and asymptomatic community-based adults with little or no advanced disease.

By integrating approaches from the physical, biological, computational, statistical and clinical sciences, this observational study will test the hypothesis that early diagnosis of subclinical signatures of critical illness encoded within physiological signals complements conventional clinical predictors by providing unique prognostic insight.

The primary goal is to reduce mortality, morbidity and complications by early identification of individuals with brewing subclinical critical illness and adverse events before overt clinical presentation (e.g., cardiac arrest, arrhythmias, hemorrhage, respiratory failure, circulatory collapse). This will provide the necessary lead time for healthcare providers to deliver early, more effective and/or preventive therapies. Through innovative approaches, CHAOS also meets the challenge of medical errors to reduce missed diagnosis, misdiagnosis, preventable harm and variability in provider adherence to best practice guidelines.

The goal is to validate predictive algorithms and identify subclinical signatures of illness, ranging from asymptomatic adults in the community to very sick patients in the hospital. The overall goal is to make healthcare more precise, effective, efficient, safe and timely while reducing costs, preventable harms and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18-100 years admitted to a bed or OR with telemetry monitoring capability will be included.

Exclusion Criteria:

* Children (individuals <18 years of age).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the hospital, including ward bed or surgical operating room with telemetry monitoring capability.
Sampling Method: Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to Mortality | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Duration of ICU/hospital stay | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

SECONDARY OUTCOMES:
Rates of critical care transfer | through study completion, an average of 1 year
Non-fatal adverse events | through study completion, an average of 1 year
readmission to unit or hospital | 30 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Cincinnati, Cincinnati, Ohio